CLINICAL TRIAL: NCT02790255
Title: BRown Fat Activity Measurement With Infrared imaginG tHermography and Thermogenesis - the BRIGHT Study
Brief Title: BRown Fat Activity Measurement With Infrared imaginG tHermography andThermogenesis - the BRIGHT Study
Acronym: BRIGHT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Singapore Institute of Food and Biotechnology Innovation (Other Government)
Collaborators: Institute for Infocomm Research (Other)
Responsible Party: Principal Investigator, Melvin Leow, Principal Investigator, Singapore Institute of Food and Biotechnology Innovation
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: 2014/00721
Record Dates: First submitted 2016-05-31; First posted 2016-06-03 (Estimated); Last update posted 2019-05-15 (Actual); Status verified 2019-05

CONDITIONS: Energy Expenditure; Obesity; Adipose Tissue, Brown
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Cold air (Experimental): Subjects to be seated in an airtight chamber at an ambient temperature between 16 to 20 degrees Celsius for 1 hour.
  Interventions: Other: Cold air
- Cold water (Experimental): Subjects to be seated in an airtight chamber at an ambient temperature of 24 degrees Celsius, with their hands and feet fully immersed in cold water for 5 minutes.
  Interventions: Other: Cold water

INTERVENTIONS:
Other: Cold air
  Arms: Cold air
Other: Cold water
  Arms: Cold water

SUMMARY:
The whole body calorimeter is sensitive enough to reliably measure cold-induced thermogenesis as a surrogate marker of brown adipose tissue (BAT) activation.

The infrared (IR) energy flux from activated BAT can be accurately imaged and quantified using an IR imaging device, and that this IR energy output may be correlated to the increased energy expenditure quantified by the whole body calorimeter.

DETAILED DESCRIPTION:
The recent rediscovery of functional brown adipose tissue (BAT) in healthy adults has opened up the exciting possibility of manipulating BAT for obesity management, and it is imperative to develop BAT imaging modalities that are non-invasive and safe for repeated use. Given that heat is a specific end-product of uncoupling protein-1 (UCP-1)-mediated BAT, this study examines whether surface body temperature assessed using infrared (IR) thermography can be a non-invasive measure to accurately and precisely predict brown adipose tissue (BAT) activation upon cold stimulation, which involves verifying an semi-automated method for characterizing thermal images. In addition, this study also aims to validate the use of a whole-body calorimeter to pick up changes in energy expenditure upon cold-induced thermogenesis. Lean, healthy male volunteers will be recruited. Thermal imaging of cervical-supraclavicular BAT will be done using an IR camera to assess changes in BAT activation. Blood samples will also be drawn at regular intervals to track changes in serum metabolites upon BAT activation. All in all, this study hopes to provide more supporting evidence that IR thermography is a viable imaging modality that is non-invasive, safe and reproducible of studying BAT activity.

ELIGIBILITY:
Inclusion Criteria:

* Male
* Ethnic Chinese
* Age between 21 to 35 years
* Body Mass Index 18.5 to 22.9
* Normal resting blood pressure ~120/80 mmHg
* Normal fasting blood glucose level <5.5 mmol/L

Exclusion Criteria:

* Do not train for or partake in competitive sports
* Do not have any major diseases
* Not on any prescribed medication

Ages: 21 Years to 35 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2014-11; Primary Completion 2018-11-05 (Actual); Study Completion 2018-11-05 (Actual)

PRIMARY OUTCOMES:
Temperature at cervical-supraclavicular region | 45 minutes cold exposure
  The temperature at the cervical-supraclavicular region following cold exposure will be determined using infrared thermal imaging.

SECONDARY OUTCOMES:
Energy expenditure during cold exposure | 45 minutes cold exposure
  Energy expenditure during cold exposure will be determined using the whole-body calorimeter.